CLINICAL TRIAL: NCT05550558
Title: Camrelizumab Plus Anlotinib in Patients With Recurrent Sporadic Mismatch Repair Deficient Endometrial Cancer (CAN-RESPOND): a Single-arm, Multicentre, Phase 2 Study
Brief Title: Camrelizumab Plus Anlotinib in Patients With Recurrent Sporadic MMRd Endometrial Cancer
Acronym: CAN-RESPOND
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-111
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-04

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — anlotinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib + Camrelizumab (Experimental): Anlotinib 12 mg QD p.o for 2 weeks and then stop for 1 week plus Camrelizumab 200 mg (fixed dose) IV every 3 weeks (+/- 3 days) until progression or adverse effects prohibit therapy
  Interventions: Drug: Anlotinib + Camrelizumab

INTERVENTIONS:
Drug: Anlotinib + Camrelizumab — Anlotinib PO plus Camrelizumab IV

SUMMARY:
Patients with advanced mismatch repair-deficient (MMRd) or microsatellite instability-high (MSI-H) endometrial cancer (EC) are currently treated as one entity, and immune checkpoint inhibitor (ICI) monotherapy is the treatment of choice. However, different molecular mechanisms drive the development of dMMR/MSI-H tumors, including germline mutations in canonical MMR genes (Lynch syndrome), somatically acquired MMR gene mutations (Lynch-like), and homozygous methylation of the MLH1 gene promoter (sporadic). There is increasing evidence that patients with sporadic MMRd EC have a worse response to ICI monotherapy than those with Lynch/Lynch-like tumors. Antiangiogenic therapy can relieve immunosuppression through blood vessel normalization and the oxygen metabolism pathway, thereby having a synergistic effect with ICIs. Anlotinib is an oral anti-angiogenic tyrosine kinase inhibitor (TKI). Camrelizumab is a fully humanized, high-affinity monoclonal antibody against PD-1. The purpose of this trial is to assess the efficacy and safety and tolerability of anlotinib plus camrelizumab in recurrent EC patients with sporadic MMRd tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must receive have completed at least 1 but no more than 3 prior lines of therapy including at least one prior platinum-based chemotherapy:

   * Patients with recurrent endometrial cancer that has failed at least one line of platinum-based chemotherapy;
   * Patients with newly diagnosed advanced (metastatic and/or unresectable) disease has persist lesion after frontline treatment with surgery and platinum-based chemotherapy ± radiotherapy;
   * Patients with newly diagnosed advanced disease that is not amenable to curative treatment with surgery and/or radiation therapy cannot tolerate chemotherapy;
2. Patients may have received prior hormonal therapy for treatment of endometrial carcinoma. All hormonal therapy must be discontinued at least one week prior to the first date of study therapy.
3. Histologically proven diagnosis of endometrial cancer.
4. Tumors must demonstrate MMRd and MLH1 methylation.

   ° Endometrial tumor MMR and MLH1 methylation status: All participants must be screened using Immunohistochemistry (IHC) for MMR proteins MLH1, MSH2, MSH6, and PMS2. MLH1 gene promoter methylation is performed in tumors exhibiting MLH1 and/or PMS2 IHC loss. MLH1 methylation status is determined by the bisulfite mediated detection of methylated cytosines, as described by Benhamida (Benhamida JK, et al. Reliable Clinical MLH1 Promoter Hypermethylation Assessment Using a High-Throughput Genome-Wide Methylation Array Platform. J Mol Diagn. 2020 Mar;22:368-375. doi: 10.1016/j.jmoldx.2019.11.005).
5. All patients must have measurable disease by RECIST 1.1.
6. ECOG performance status 0-2.
7. Life expectancy ≥ 12 weeks.
8. Patients must have adequate organ function:

   * Absolute neutrophil count (ANC) ≥ 1.5×10^9/L;
   * Platelet count ≥ 70 × 10^9/L;
   * Hemoglobin ≥ 80 g/L;
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN);
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN (however, patients with known liver metastasis who have AST or ALT level ≤ 5 × ULN may be enrolled);
   * Creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula);
   * Baseline albumin ≥ 25 g/L;
   * Thyroid-stimulating hormone (TSH) levels ≤ 1 × ULN (however, patients with free Triiodothyronine [FT3] or free Thyroxine [FT4] levels ≤ 1 × ULN may be enrolled)
9. Signed and dated informed consent.

Exclusion Criteria:

1. Histologically confirmed diagnosis of sarcoma components including malignant mixed mullerian tumors.
2. Patients who have had prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune check point pathways.
3. History of severe hypersensitivity reaction (≥Grade 3) to any monoclonal antibody.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure and unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Uncontrolled hypertension (blood pressure >140/90 mmHg) after adequate treatment.
6. Central nervous system diseases, including uncontrollable epilepsy and central nervous system metastases.
7. Radiographically confirmed major blood vessel invasion/infiltration.
8. Prior chemotherapy, targeted small molecule therapy, bevacizumab, or radiation therapy within 4 weeks of study Day 1 or not recovered from adverse events caused by previously administered treatment.
9. Prior hormonal therapy for the treatment of endometrial carcinoma within 1 weeks of study Day 1.
10. Known history of Human Immunodeficiency Virus (HIV).
11. Known active tuberculosis (TB, Bacillus tuberculosis).
12. Known active Hepatitis B or C.
13. known active ulcer, or active colitis.
14. Received live vaccine within 30 days of planned start of study treatment.
15. Patients who have gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of anlotinib.
16. Patients who have severe gastrointestinal or non-gastrointestinal fistula (≥Grade 3).
17. Patients who have an allogenic tissue/solid organ transplant.
18. Patients who have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

    ⁕⁕⁕Note:
    * Topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption) are permitted;
    * Physiologic replacement doses of systemic corticosteroids are permitted, even if <10 mg/day prednisone equivalents are permitted;
    * A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted;
19. Is pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Frequency and severity of adverse events (AEs) | 24 months
  Number of participants with AEs occurring up to 28 days after the last administration are evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03.
Progression-free Survival (PFS) | 24 months
  The duration from date of enrollment to the disease progression, death, or the date of last contact, whichever occurs first.
Overall Survival (OS) | 24 months
  The duration from date of enrollment to time of death or the date of last contact, , whichever occurs first.
Disease Control Rate (DCR) | 24 months
  The percentage of participants in the analysis population who have a CR, PR or SD as assessed by RECIST 1.1.
Duration of Response (DOR) | 24 months
  the time from first documented CR or PR until disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Yan-fang Ye, PhD, Study Director — Clinical Research Design Division, Sun Yat-sen Memorial Hospital

IPD SHARING:
Plan to Share IPD: Yes
The protocol and statistical analysis plan will be made available on Clinicaltrials.gov.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: email lijing228@mail.sysu.edu.cn